CLINICAL TRIAL: NCT06712511
Title: The Effect of Coffee on Energy Expenditure and Caffeine Metabolism
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences (Other)
Responsible Party: Principal Investigator, John R. Speakman, Professor, Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: SIAT IRB 240715H0902
Record Dates: First submitted 2024-11-26; First posted 2024-12-02 (Actual); Last update posted 2025-03-27 (Actual); Status verified 2025-03

CONDITIONS: Healthy
Keywords: Coffee; Caffeine; Energy expenditure; Caffeine metabolism

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- water (Experimental): The participants will drink 200 ml water four times at 1 hour intervals.
  Interventions: Other: Caffeine content
- coffee (Experimental): The participants will drink 200 ml coffee four times at 1 hour intervals.
  Interventions: Other: Caffeine content

INTERVENTIONS:
Other: Caffeine content — Participants will drink the same volume of water or coffee, caffeine content is 2mg/kg by body weight.

SUMMARY:
Obesity is a risk factor for chronic diseases, and improving energy expenditure is a way to prevent and treat obesity. The purpose of this project is to explore the relationship between the effect of coffee on energy expenditure and caffeine metabolism, which has important significance in the rational application of caffeine.

DETAILED DESCRIPTION:
The investigators will study the relationship between the effect of coffee on energy expenditure and caffeine metabolism. The investigators will recruit healthy participants. Participants will be forbidden to consume stimulant drinks such as coffee for 24 hours before the experiment. When the participants arrive at the lab on the day of the experiment, they will sign an informed consent form, a health history questionnaire and a daily coffee consumption questionnaire. The changes of drinking water/coffee on total energy expenditure (TEE), body temperature, heart rate, blood pressure, electrocardiogram, memory，cognition, sleep time and so on will be observed. The concentration of caffeine and its metabolites in the blood and urine will be measured by liquid chromatography-mass spectrometry (LC-MS) and gas chromatography-mass spectrometry (GC-MS).

ELIGIBILITY:
Inclusion Criteria：

* Healthy adults.
* Must be able to drink coffee.

Exclusion Criteria:

* Diabetes.
* Hypoglycemia.
* Gout.
* Osteoporosis.
* Gastric ulcer.
* Pancreatitis.
* Intestinal obstruction.
* Blood phobia.
* Pathological hypo or hyper tension.
* Impaired glucose tolerance.
* Claustrophobia.
* HIV,etc.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2024-10-23 (Actual); Primary Completion 2029-06-30 (Estimated); Study Completion 2029-12-31 (Estimated)

PRIMARY OUTCOMES:
Total energy expenditure | 2 days
  Total energy expenditure will be measured by Chamber (OMNICAL).
The concentration of caffeine and its metabolites in urine | 2 days
  The contents of caffeine and it's metabolites will be measured by gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS ).
The concentration of caffeine and its metabolites in serum | 1 day
  The concentration of caffeine and its metabolites in serum will be measured by gas chromatography-mass spectrometry (GC-MS) and liquid chromatography-mass spectrometry (LC-MS ).

SECONDARY OUTCOMES:
Body temperature | 2 days
  Body temperature of participants will be measured by body temperature patch (RIT-P02-MED).
Electrocardiogram (ECG) | 2 days
  ECG of participants will be measured by Amu ECG belt, the changes in P wave, PR interval, PR segment, QRS wave group, J point, ST segment, T wave, QT interval, and U wave will be observe.
Blood pressure | 2 days
  Systolic and diastolic blood pressure of participants will be measured by Omron digital sphygmomanometer.
Height | The morning of the first day of the experiment, 5 mins
  Height will be measured by seca 217 stable stadiometer. Subjects wearing no shoes.
Body weight | The morning of the first day of the experiment, 5 mins
  Fasting body weight will be measured by Bioimpedance Analysis (TANITA, MC-980).
Fat mass | The morning of the first day of the experiment, 10 mins
  Fat mass will be measured by Magnetic Resonance Imaging (Shanghai united imaging, uMR 790 ).
Fat free mass | on the morning of the experiment, 5 mins
  Fat free mass will be Bioimpedance Analysis (Tanita, MC-980).
Heart rate | 2 days
  Heart rate will be measured by Polar heart rate belts.
Hunger rating | 2 days
  Hunger score will be measured on (Visual Analogue Scale) VAS by a pen and a paper. According to the scores of each participant, the highest score was 100 % hunger rate, and hunger rate (%) at other time points will be obtained from hunger score × 100 % / the highest score.
Memory and cognitive tests | The morning of the experiment, 60 mins
  Memory and cognitive tests will be tested by Cognitive Experiment Standard Toolbox (CEST).
Physical activity | 7 days
  The physical activity of volunteers will be recorded by accelerometer (GT3XP-BTLE).
Sleep duration | 2 days
  The sleep duration of volunteers will be recorded by polar watch.
Waist circumferences | The morning of the first day of the experiment,10 mins.
  Waist circumferences will be measured using a whole body laser scanner (TG2000-F).

CONTACTS AND LOCATIONS:
Overall Officials: John R Speakman, PhD, Study Chair — Shenzhen Institutes of Advanced Technology ,Chinese Academy of Sciences
Locations (1):
- Shenzhen Institute of Advanced Technology, Chinese Academy of Sciences, Shenzhen, Guangdong, China